CLINICAL TRIAL: NCT01478698
Title: A Phase 1, Open Label, Non Randomised Safety Trial of Intraperitoneal tPA and DNase in Peritoneal Dialysis Patients With Peritonitis
Brief Title: The Safety and Tolerability of Intra-abdominal t-PA and DNase on Peritonitis in Peritoneal Dialysis Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient budget for further study agents
Sponsor: Sir Charles Gairdner Hospital (Other)
Collaborators: The University of Western Australia (Other)
Responsible Party: Principal Investigator, Aron Chakera, Dr, Sir Charles Gairdner Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tPADNase 1
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Peritoneal Dialysis; Peritoneal Dialysis, Continuous Ambulatory
Keywords: peritoneal dialysis; peritoneal dialysis, continuous ambulatory; peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Tissue Plasminogen Activator; dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single dose (Experimental): The first 5 consented participants will be administered t-PA 10mg + DNase 5mg instilled into a dialysate bag and infused for a 4 hour intraperitoneal dwell.
  Interventions: Drug: Tissue Plasminogen Activator (tPA); Drug: recombinant deoxyribonuclease (DNase)
- 2 doses (Experimental): The next 5 consented participants will be administered t-PA 10mg + DNase 5mg instilled twice a day for one day
  Interventions: Drug: Tissue Plasminogen Activator (tPA); Drug: recombinant deoxyribonuclease (DNase)
- 4 doses (Experimental): The next 5 consented participants will be administered tPA 10mg + DNase 5mg twice a day for 2 days.
  Interventions: Drug: Tissue Plasminogen Activator (tPA); Drug: recombinant deoxyribonuclease (DNase)
- control (No Intervention): Any potential participants that have not consented into the intervention arms will be approached to be consented into a non-intervention observational control group. A maximum of 5 participants will be recruited into this control group.

INTERVENTIONS:
Drug: Tissue Plasminogen Activator (tPA) — tPA 10mg per dose intraperitoneal
  Arms: 2 doses; 4 doses; Single dose
Drug: recombinant deoxyribonuclease (DNase) — DNase 5mg per dose given intraperitoneally.
  Arms: 2 doses; 4 doses; Single dose

SUMMARY:
Hypothesis:

Intraperitoneal tPA and DNase is well tolerated at a number of different doses. Different doses of tPA and DNase will have a dose-related effect on inflammatory markers (CRP and intraperitoneal white cell count).

Aims:

1. To examine the tolerability of different doses of intraperitoneal tPA and DNase compared to standard treatment.
2. To examine the changes in biochemical and clinical outcomes of PD Peritonitis with the addition of intraperitoneal tPA and DNase to usual therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PD patient
2. Proven peritonitis (as defined as at least 2 of: (i) Symptoms and/or signs of peritonitis; (ii) Cloudy dialysate OR dialysate white cell count > 100x 106/L with >50% neutrophils; (iii) Positive culture of dialysate
3. Age > 18 years old

Exclusion Criteria:

1. More than one organism on culture
2. Contra-indication for systemic thrombolysis (eg. current or recent stroke, major haemorrhage or major trauma; proliferative retinopathy; major surgery in the previous 5 days)
3. Known sensitivity to DNase or t-PA
4. Pregnancy or lactating mother
5. Expected survival less than 3 months
6. Clinical indication for PD catheter removal, as defined by treating team
7. Inability to provide written informed consent
8. Systemic anticoagulation
9. Severe uncontrolled hypertension
10. Documented ulcerative gastrointestinal disease during the last three months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Adverse reactions | 72 hours
  Participants will be examined for potential adverse reactions during this trial, including - pain; abnormalities in systemic coagulation profile; bleeding; and altered blood pressure.

SECONDARY OUTCOMES:
Biochemical markers of inflammation | 21 days
  Biochemical markers of inflammation will be measured on days 1, 3, 5, 7, 14 and 21, including - c-reactive protein, white cell count, dialysate white cell count, procalcitonin
Clinical markers of inflammation | 21 days
  pain score; days till pain free; proportion requiring catheter removal; days of hospitalisation; days of fever (temperature > 37.0 degrees on at least one occasion)

OTHER OUTCOMES:
Additional variables | 3 months
  gentamycin and vancomycin levels, ultrafiltration volume; mortality; relapse and recurrence rates of peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Aron Chakera, DPhil, Study Director — Sir Charles Gairdner Hospital
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia